CLINICAL TRIAL: NCT06587516
Title: Developing a Novel Neuromuscular Warm-Up Program for Recreational Badminton Players: An Experimental Study
Brief Title: Neuromuscular Warm-Up Program for Badminton Players
Acronym: NWUPFBM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Saranya Navaratnarajah, Ms, University of Malaya
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: UM.TNC2/UMREC_3398
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Balance; Distorted; Ankle Injury
Keywords: Recreational Badminton; Balance Improvement; Ankle Injury Prevention; Neuromuscular Warm Up; Warm Up Program
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Intervention Model Description: This study uses a crossover design where each participant will experience both the neuromuscular warm-up program (intervention) and the traditional warm-up (control). The order of the interventions will be randomized. After completing the first condition, participants will have a one-day washout period before switching to the other condition. This design allows each participant to serve as their own control, which enhances the comparison between the effects of the two conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): badminton players who plays badminton socially once a week with minimum experience of three years
  Interventions: Behavioral: Neuromuscular Warmup Program
- Control (Active Comparator): badminton players who plays badminton socially once a week with minimum experience of three years
  Interventions: Behavioral: Traditional Warmup Program

INTERVENTIONS:
Behavioral: Neuromuscular Warmup Program — This intervention consists of a structured warm-up routine specifically designed to enhance neuromuscular function and balance. The program includes exercises such as two way forward lunge, single-leg balance, multidirectional lunges, single-leg hops forward and backward, and single-leg calf raises. Each exercise is aimed at improving proprioception, dynamic stability, and lower limb strength.
  Arms: Experimental
Behavioral: Traditional Warmup Program — This intervention involves a conventional warm-up program. It includes general stretching exercises and light jogging intended to prepare the body for physical activity.
  Arms: Control

SUMMARY:
This study aims to develop and evaluate a new warm-up program specifically designed for recreational badminton players. The program focuses on exercises that enhance balance and reduce the risk of ankle injury. Participants will be asked to follow this warm-up routine, and their performance will be assessed before and after to see if the exercises improve their balance and overall movement. The goal is to create a practical, effective warm-up routine that can be easily incorporated into badminton practice.

DETAILED DESCRIPTION:
This study investigates the effectiveness of a novel neuromuscular warm-up program tailored for recreational badminton players. The program is designed to improve balance, enhance movement efficiency and reduce the risk of injuries commonly associated with badminton.

Participants will be recruited from recreational badminton clubs and will undergo baseline assessments of balance performance and lunge movement using motion capture (Mocap), EMG. and inertia measurement unit (IMU). The warm-up program includes a series of targeted exercises selected based on expert consensus from a previous Delphi study. These exercises focus on key areas such as dynamic stability, and proprioception.

Participants perform pre and post test with Star Excursion Balance Test (SEBT) and forward lunge movement with (IMU, MOcap and MEG) attached on the lower limb. The intervention will be: 1) novel neuromuscular warmup and 2) traditional warmup. Participants will perform both the warmup but on different days with one day rest in between the interventions.

The study's findings aim to inform best practices for warm-up routines in badminton, potentially offering a standardized program that can be widely adopted by recreational players to enhance their performance and safety on the court.

ELIGIBILITY:
Inclusion Criteria:

* Injury free for >1 year, plays badminton minimum of once a week, have experience of playing at least 3 years

Exclusion Criteria:

* Badminton players that participate in competition in any level (novice, intermediate or elite tier), involve in any regimented training, participants with any joint disorder, non-communicable diseases (NCD), neurologically unstable, consumption of any medication that can interfere with performance.

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
Balance Performance | pre-test conducted immediately before the intervention and a post-test conducted immediately after the intervention
  Balance will be measured using standardised tests such as the Star Excursion Balance Test (SEBT), which evaluates the participant's reach distances in multiple directions
Ankle Movement | pre-test conducted immediately before the intervention and a post-test conducted immediately after the intervention.
  This measure will assess the angle of (dorsi-flexion and plantar-flexion) and (inversion and eversion) at the ankle joint during the lunge movement. The aim is to evaluate changes in ankle joint alignment and range of motion as a result of the neuromuscular warm-up program. Ankle angles will be measured using motion capture technology and an inertial measurement unit (IMU) to provide accurate and objective data.

SECONDARY OUTCOMES:
Neuromuscular Activity | pre-test conducted immediately before the intervention and a post-test conducted immediately after the intervention
  This measure will evaluate neuromuscular activity using electromyography (EMG) to assess muscle activation patterns during the lunge movement. EMG sensors will be placed on key muscles involved in the lunge, such as the quadriceps, hamstrings, and calf muscles, to record electrical activity. This data will help determine the impact of the neuromuscular warm-up program on muscle activation, coordination, and overall neuromuscular function during dynamic movements.

CONTACTS AND LOCATIONS:
Overall Officials: Saranya Navaratnarajah, Principal Investigator — Institute for Advanced Studies, Universiti Malaya
Locations (1):
- University of Malaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Akbari M, Karimi H, Farahini H, Faghihzadeh S. Balance problems after unilateral lateral ankle sprains. J Rehabil Res Dev. 2006 Nov-Dec;43(7):819-24. doi: 10.1682/jrrd.2006.01.0001. PMID 17436168